CLINICAL TRIAL: NCT00847587
Title: Randomized Controlled Trial of Early Versus Standard Postpartum Insertion of the Etonogestrel Contraceptive Implant
Brief Title: Early Versus Standard Postpartum Insertion of the Etonogestrel Contraceptive Implant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, David Turok, M.D., University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30291
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Results first posted 2011-06-02 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-03

CONDITIONS: Complications; Contraceptive; Female Lactation
Keywords: Contraceptive; Implant; Postpartum period; etonogestrel-releasing; lactogenesis; Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Early postpartum insertion
  Interventions: Drug: Etonogestrel contraceptive implant
- 2 (Active Comparator): Standard postpartum insertion
  Interventions: Drug: Etonogestrel contraceptive implant

INTERVENTIONS:
Drug: Etonogestrel contraceptive implant — Implant insertion postpartum prior to hospital discharge
  Arms: 1
Drug: Etonogestrel contraceptive implant — Standard insertion at 4-8 weeks postpartum
  Arms: 2

SUMMARY:
A highly effective single rod contraceptive implant is now available for use in the US. Delays in the insertion of the device until later in the postpartum period may negatively impact initiation rates. The objective of this study is to compare outcomes of early postpartum insertion (prior to postpartum hospital discharge) of the etonogestrel-releasing contraceptive implant with routine postpartum insertion at 4-8 weeks after delivery. Primary outcome of interest will be time to lactogenesis. Secondary outcomes will include rates of breastfeeding supplementation, infant growth, vaginal bleeding patterns, incidence of side effects, time to resume sexual intercourse after delivery, and incidence of missed routine postpartum follow-up. In addition, a subset of patients who randomize to early postpartum insertion will have expressed breastmilk ascertained for nutrient composition.

DETAILED DESCRIPTION:
This is a randomized controlled trial. Participants will be assigned with equal probability to 1 of the 2 test groups using computer-generated random numbers in blocks of varying sizes. Allocation concealment will be assured by enclosing assignments in sequentially numbered, opaque, sealed envelopes. Envelopes will be opened sequentially and only after the participant's name and study number are written on the envelope. Follow-up and data collection for participants in each group will be identical. Outcome assessors and data analysts will be blinded to treatment arm.

STUDY PROCEDURES:

Inclusion/exclusion criteria will be verified and consent obtained. The patient will be notified of the results of randomization and the physician able to perform insertion will be contacted to perform the insertion. All insertions will be performed by physicians who have completed Implanon® insertion training. If the patient randomizes to standard postpartum insertion, she will be given a clinic appointment in 4-8 weeks for the insertion procedure.

Lactogenesis time will be documented by maternal perception, as described and validated by Chapman et al16. If lactogenesis has not occurred prior to hospital discharge, the patient will receive daily phone calls from study personnel until lactogenesis can be confirmed and recorded. Contact information for the patient, as well as for two friends or relatives who will know how to reach her will be obtained and verified prior to discharge. Participants will be given a reminder card for the telephone calls from the investigator and a postpartum visit appointment. Patients will be instructed to contact the investigators immediately for pain, excessive bleeding, difficulty with breastfeeding, or other concerns. Patients will be given a log book ("diary") to record breastfeeding parameters including use of supplementation, infant weights, side effects, return to sexual intercourse, contraceptive method use, and days of bleeding for the study follow-up period.

Clinical follow-up will be as follows. Postpartum telephone calls or visits to collect additional data will occur as needed for up to 5 days following hospital discharge, at 2 weeks, 4-8 weeks, and 3 and 6 months postpartum. Information obtained at these points will include: breastfeeding status and parameters, collection of record of infant weights (birth, 4-8 weeks, and 6 months), reminders to keep weekly diary, collection of diaries (6 month visit), resumption of sexual activity, use of contraceptive method, and satisfaction with contraceptive method. Patients randomized to early insertion will be asked to give a milk sample for analysis at their 4-8 week visit. Table 1 describes the contact points with the subject for collection of data. Contact will be either by telephone or at clinic visits.

ELIGIBILITY:
Inclusion Criteria: Patients on the postpartum ward at University Hospital will be offered inclusion in the study if they are:

* healthy,
* 18-40 years old,
* delivered a healthy term infant,
* intend to breastfeed,
* desire Implanon as their method of contraception, and
* agree to be randomized to early versus standard postpartum insertion.

Exclusion Criteria:

* obstetric complications including anemia with hematocrit<30,
* transfusion,
* infection,
* severe pregnancy induced hypertension,
* prolonged hospitalization,
* coagulopathy,
* liver disease,
* undiagnosed genital bleeding,
* or other relative contraindication to Implanon® insertion (known or suspected pregnancy, known, suspected, or history of breast cancer, or hypersensitivity to any of the components in Implanon®).
* Women taking drugs that are potent inducers of hepatic enzymes will also be excluded, including barbiturates, griseofulvin, rifampin, phenylbutazone, phenytoin, carbamazepine, felbamate, oxcarbazepine, topiramate, modafinil, protease inhibitors, and herbal products including St. John's Wort.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shawn E Gurtcheff, MD, Principal Investigator — University of Utah; David K Turok, MD, Study Chair — University of Utah; Kirtly P Jones, MD, Study Director — University of Utah; Patricia Murphy, DrPH, Study Director — University of Utah; Sara E Simonsen, RN, BSN, Study Director — University of Utah
Locations (1):
- University of Utah Hospital, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Gurtcheff SE, Turok DK, Stoddard G, Murphy PA, Gibson M, Jones KP. Lactogenesis after early postpartum use of the contraceptive implant: a randomized controlled trial. Obstet Gynecol. 2011 May;117(5):1114-1121. doi: 10.1097/AOG.0b013e3182165ee8. PMID 21508750

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in the postpartum ward of the University of Utah hospital. Recruitment took place during 2009-2010.
Pre-assignment Details: Randomization occurred after consent. No participants were excluded from the trial after randomization.
Groups:
- Early Postpartum Insertion: Early postpartum insertion of the etonogestrel contraceptive implant: insertion performed by the third postpartum day.
- Standard Postpartum Insertion: Standard postpartum insertion of the etonogestrel contraceptive implant: insertion performed at 4-8 weeks postpartum.
Period: Overall Study
Arm/Group | Early Postpartum Insertion | Standard Postpartum Insertion
Started | 35 | 34
Completed | 34 (Patient declined study after randomization.) | 34
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Postpartum Insertion | Standard Postpartum Insertion | Total
Number analyzed (Participants) | 35 | 34 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (6) | 25 (6) | 26 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 34 | 69
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 34 | 69

OUTCOME MEASURES:

1. Primary Outcome: Time to Lactogenesis Stage II
Description: The primary outcome, time to lactogenesis stage II in hours, was documented by maternal perception as previously described and validated in the literature. Subjects were asked, "Has your milk come in? Some women experience this as a prickly feeling or tingling in the breast, dripping from the other nipple when nursing, milk running from the baby's mouth, or gulping by the baby. " If the response was positive, subjects were then asked, "When did your milk come in?" and the response recorded to the nearest hour.
Time Frame: 5 days postpartum
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Early Postpartum Insertion | Standard Postpartum Insertion
Number analyzed (Participants) | 35 | 34
hours | 64.3 (19.6) | 65.2 (18.2)
Statistical Analysis 1: Comparison: Early Postpartum Insertion vs Standard Postpartum Insertion; It was assumed that both groups would have a mean of 54 hours to lactogenesis with a common standard deviation of 12 hours based on previous reports of lactogenesis in women with uncomplicated vaginal deliveries. Setting the noninferiority margin at 8 additional hours, using an alpha 0.05 level comparison, to achieve 80% power a sample size of n=34 evaluable subjects was required in each group. The calculation was performed using N Solution 2007 Professional Software; Test type: Non-Inferiority or Equivalence — A noninferiority margin of 8 additional hours was chosen to be clinically relevant, as many common medical interventions (such as epidural anesthesia, cesarean delivery, labor induction, and general stress) have been reported to delay time to lactogenesis stage II by up to 12 hours; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-10.6 to 7.7], Standard Deviation 120

2. Secondary Outcome: Crematocrit of Human Milk
Description: Determination of creamatocrit is a simple method for estimating the fat & energy content of human milk based on the centrifugation of milk in a hematocrit centrifuge. The method for creamatocrit measurement was as described by Lucas et al (LucasA, GibbsJA, LysterRL, BaumJD. Creamatocrit: simple clinical technique for estimating fat concentration and energy value of human milk. BritMedJnl1978;1:1018-20)using a standard hematocrit centrifuge, standard hematocrit glass capillary tube, & vernier calipers. Measurements were performed in duplicate and the mean for each measurement used for analysis.
Time Frame: 6 weeks postpartum
Population: Both intent-to-treat and per-protocol analyses were performed. Per-protocol analysis is presented to demonstrate the more conservative analysis for the primary outcomes in a noninferiority study.
Measure: Mean (Standard Deviation); unit: Percent creamatocrit
Arm/Group | Early Postpartum Insertion | Standard Postpartum Insertion
Number analyzed (Participants) | 21 | 22
Percent creamatocrit | 7.5 (3) | 6.8 (3.2)
Statistical Analysis 1: Comparison: Early Postpartum Insertion vs Standard Postpartum Insertion; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Risk Difference (RD) = 0.61, 95% CI 2-sided [-1.3 to 2.5], Standard Deviation 1.8

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 6 months from delivery.
Arm/Group | Early Postpartum Insertion | Standard Postpartum Insertion
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/34
Other Adverse Events (participants affected / at risk) | 0/35 | 0/34

LIMITATIONS AND CAVEATS:
Limitations:Study was not blinded & early insertion was allowed as late as 3 days postpartum. Insertion on postpartum days 1-3 was allowed so long as lactogenesis had not already occurred to mimic normal clinical practice & improve generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No